CLINICAL TRIAL: NCT05878223
Title: The Dose Effectiveness of Extracorporeal Shockwave on Plantar Flexor Spasticity of Ankle in Stroke Patients: a Randomised Controlled Trial
Brief Title: Comparing ESWT Doses for Post-Stroke Ankle Spasticity Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital Hsin-Chu Branch (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111-044-F
Record Dates: First submitted 2023-01-03; First posted 2023-05-26 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Stroke
Keywords: stroke; spasticity; shock wave; ankle
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESWT to gastrocnemius and soleus (Experimental): ESWT to gastrocnemius and soleus muscles (2000 shots for each muscle, a total of 4000 shots per session)
  Interventions: Device: Extracorporeal shock waves
- ESWT to gastrocnemius (Active Comparator): ESWT to gastrocnemius muscle (2000 shots per session)
  Interventions: Device: Extracorporeal shock waves

INTERVENTIONS:
Device: Extracorporeal shock waves — Both group received extracorporeal shock waves therapy

SUMMARY:
Post-stroke spasticity is a common complication affecting the neurological recovery, self-care daily activities and patients' quality of life. Extracorporeal shock waves (ESWT) have been proven therapeutic effects on decreasing spasticity and regaining function. Stroke patients often suffer ankle plantar flexor spasticity with poor ankle movement control, leading to abnormal gait patterns and risk of falling; local pain appears as well in the ankle. Research showed application of ESWT to lower extremity spasticity reduced ankle plantar flexor spasticity, ankle pain and increased the range of ankle motion. However, the current study did not investigate the effect of ESWT on different muscles in patients with post-stroke ankle spasticity. Therefore, this study will compare the effect of focused ESWT on combination of the gastrocnemius and soleus muscles to gastrocnemius muscle alone in the post-stroke ankle plantar flexor spasticity.

DETAILED DESCRIPTION:
This study design was a single-blind randomized controlled trial and planned to recruit 40 chronic stroke patients with ankle plantar flexor spasticity. The patients were randomly assigned to two groups. The experimental group received focused ESWT to gastrocnemius and soleus muscles (a total of 4000 shots per session), while the control group received focused ESWT to gastrocnemius muscle (2000 shots per session). Patients in both groups underwent a total of 4 sessions ESWT, twice a week for two consecutive weeks. The primary outcome was modified Ashworth scale; the secondary outcomes were modified Tardieu scale, passive range of ankle motions and timed up and go test, and strain elastography. The outcomes were assessed before ESWT and after ESWT at 1, 4, 12, and 24 week.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with Cerebral stroke and age more 20
2. The degree of spasticity of plantar flexor is more than 1.( grading with the modified Ashworth scale)
3. Stable vital sign

Exclusion Criteria:

1. Recurrent cerebral stroke, traumatic brain injury, brain tumor or other brain related disease.
2. Other central nervous system diseases (SCI, Parkinson's disease), or other musculoskeletal disorders which affect the result of evaluating muscle spasticity.
3. Malignant tumor, coagulation disorder, infection or use of pace which were not suitable for Extracorporeal Shock Wave.
4. Received Extracorporeal Shock Wave or Botulinum injection for plantar flexor spasticity in recent 3 months.
5. Subjects who was unable to complete Extracorporeal Shock Wave or evaluation due to impaired cognition or aphasia.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Ashworth Scale (MAS) | T0 Enrollment, T1 after 1 week from T0, T2 after 4 weeks from T0, T3 after 12 weeks from T0, T4 after 24 weeks from T0
  Modified Ashworth Scale (MAS). Score from 0 to 4, higher scores mean a worse outcome

SECONDARY OUTCOMES:
Change in Level of mobility and balance | T0 Enrollment, T1 after 1 week from T0, T2 after 4 weeks from T0, T3 after 12 weeks from T0, T4 after 24 weeks from T0
  Timed Up & Go Test
Ultrasound evaluations | T0 Enrollment, T1 after 1 week from T0, T2 after 4 weeks from T0, T3 after 12 weeks from T0, T4 after 24 weeks from T0
  Strain elastography of gastrocnemius muscle
Barthel index | T0 Enrollment, T1 after 1 week from T0, T2 after 4 weeks from T0, T3 after 12 weeks from T0, T4 after 24 weeks from T0
  measures a person's daily living abilities, focusing on ten areas of self-care and mobility. Scores range from 0 to 100, with higher scores denoting greater independence.
Change in modified Tardieu scale (mTS) | T0 Enrollment, T1 after 1 week from T0, T2 after 4 weeks from T0, T3 after 12 weeks from T0, T4 after 24 weeks from T0
  Modified Tardieu scale (mTS). Score from 0 to 5, higher scores mean a worse outcome
Change in Passive ROM of the ankle in dorsiflexion | T0 Enrollment, T1 after 1 week from T0, T2 after 4 weeks from T0, T3 after 12 weeks from T0, T4 after 24 weeks from T0
  Passive ankle Range of Motion (PROM)

CONTACTS AND LOCATIONS:
Overall Officials: Meng Ting Lin, MD, Principal Investigator — The Department of Physical Medicine and Rehabilitation, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital Hsin-Chu Branch, Hsinchu, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ward AB. A literature review of the pathophysiology and onset of post-stroke spasticity. Eur J Neurol. 2012 Jan;19(1):21-7. doi: 10.1111/j.1468-1331.2011.03448.x. Epub 2011 Jun 27. PMID 21707868
- [Background] Mariotto S, de Prati AC, Cavalieri E, Amelio E, Marlinghaus E, Suzuki H. Extracorporeal shock wave therapy in inflammatory diseases: molecular mechanism that triggers anti-inflammatory action. Curr Med Chem. 2009;16(19):2366-72. doi: 10.2174/092986709788682119. PMID 19601786
- [Background] Yoon SH, Shin MK, Choi EJ, Kang HJ. Effective Site for the Application of Extracorporeal Shock-Wave Therapy on Spasticity in Chronic Stroke: Muscle Belly or Myotendinous Junction. Ann Rehabil Med. 2017 Aug;41(4):547-555. doi: 10.5535/arm.2017.41.4.547. Epub 2017 Aug 31. PMID 28971038
- [Background] Fan T, Zhou X, He P, Zhan X, Zheng P, Chen R, Li R, Li R, Wei M, Zhang X, Huang G. Effects of Radial Extracorporeal Shock Wave Therapy on Flexor Spasticity of the Upper Limb in Post-stroke Patients: Study Protocol for a Randomized Controlled Trial. Front Neurol. 2021 Sep 9;12:712512. doi: 10.3389/fneur.2021.712512. eCollection 2021. PMID 34566855
- [Result] Li TY, Chang CY, Chou YC, Chen LC, Chu HY, Chiang SL, Chang ST, Wu YT. Effect of Radial Shock Wave Therapy on Spasticity of the Upper Limb in Patients With Chronic Stroke: A Prospective, Randomized, Single Blind, Controlled Trial. Medicine (Baltimore). 2016 May;95(18):e3544. doi: 10.1097/MD.0000000000003544. PMID 27149465
- [Derived] Yang SM, Chen YH, Lu YL, Wu CH, Chen WS, Lin MT. The dose effectiveness of extracorporeal shockwave on plantar flexor spasticity of ankle in stroke patients: a randomized controlled trial. J Neuroeng Rehabil. 2024 Oct 1;21(1):176. doi: 10.1186/s12984-024-01473-z. PMID 39354619